CLINICAL TRIAL: NCT03157804
Title: Clinical Trial Phase I / II to Evaluate the Safety and Efficacy of the Infusion of Autologous CD34 + Cells Transduced With a Lentiviral Vector Carrying the Gene FANCA in Patients With FA Subtype A (FANCOLEN-1)
Brief Title: Lentiviral-mediated Gene Therapy of Fanconi Anemia Patients Subtype A
Acronym: FANCOLEN-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other)
Collaborators: Centro de Investigaciones Energéticas, Medioambientales y Tecnológicas (CIEMAT) (Unknown); Centro de Investigación en Red de Enfermedades Raras (CIBERER) (Unknown); Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other); Hospital Vall d'Hebron (Other); Universitat Autonoma de Barcelona (Other)
Responsible Party: Principal Investigator, Julian Sevilla, M.D.PhD Specialist in Hematology Hemotherapy, Responsible for the Transfusion Service and Unit for the Obtention and Processing of Hematopoietic Progenitors and other cellular therapies at the Hospital Infantil Universitario Niño Jesús de Madrid., Hospital Infantil Universitario Niño Jesús, Madrid, Spain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-006100-12
Record Dates: First submitted 2017-04-26; First posted 2017-05-17 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Fanconi Anemia
MeSH Terms: conditions — Fanconi Anemia | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Colony-Stimulating Factors; plerixafor; ferric pyrophosphate

ARMS (1):
- Autologous CD34+ cells transducted with PGK-FANCA-Wpre * (Experimental): CD34 + cells from patients with Fanconi subtype A (FA-A) transduced ex vivo with lentiviral vector carrying the gene FANCA, PGK-FANCA-Wpre*The product to be infused consist of a suspension of transduced CD34^+ cells.
  Interventions: Procedure: IV administration of Genetically Engineered Hematopoietic Stem/Progenitors Cells (HSPCs); Biological: Genetically Engineered Hematopoietic Stem/Progenitor Cells; Other: Laboratory Biomarker Analysis; Biological: Filgrastim; Drug: Plerixafor; Procedure: Bone Marrow Aspiration

INTERVENTIONS:
Procedure: IV administration of Genetically Engineered Hematopoietic Stem/Progenitors Cells (HSPCs)
Biological: Genetically Engineered Hematopoietic Stem/Progenitor Cells — Undergo infusion of genetically modified hematopoietic progenitor cell therapy
  Other Names: Genetically Engineered HSPCs
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Filgrastim — Given subcutaneously (SC)
  Other Names: Filgrastim XM02, Filgrastim-sndz, G-CSF (Colony Stimulating Factor), Neupogen, r-metHug-CSF, Recombinant Methionyl Human Granulocyte CSF, rG-CSF, Tbo-filgrastim, Zarxio
Drug: Plerixafor — Given SC
  Other Names: AMD 3100, JM-3100, Mozobil, SDZ SID 791
Procedure: Bone Marrow Aspiration

SUMMARY:
This is an open, Phase I / II clinical trial to evaluate the safety and efficacy of a hematopoietic gene therapy procedure with an orphan drug consisting of a lentiviral vector carrying the FANCA gene for patients with Fanconi Anemia of Subtype A .

CD34 + cells derived from bone marrow and / or mobilized peripheral blood (fresh and / or cryopreserved) from patients with Fanconi subtype A (FA-A), will be transduced ex vivo with a lentiviral vector carrying the gene FANCA (orphan drug) . After transduction the cells will be inoculated in patients in order to restore their hematopoiesis with genetically corrected stem cells.

DETAILED DESCRIPTION:
The main objective of this open-label Phase I / II clinical trial is to evaluate the safety and therapeutic efficacy of a hematopoietic gene therapy procedure with an orphan drug consisting of a lentiviral vector carrying the FANCA gene for patients with Fanconi's Anemia Subtype A.

The drug to be administered to the patients consists of the cellular product resulting from the transduction of autologous CD34 + cells with the therapeutic lentiviral vector PGK-FANCA.Wpre *.

The dose of cells to infuse in the patients will be that obtained from the transduction process of between 3x10^5 and 4x10^6 CD34 + cells / kg of patient body weight.

The cells will be infused intravenously in a single dose, after complete the transduction process.

Follow-up period: 3 years after infusion of transduced cells. However, patients will be monitored outside the clinical trial over a 10-year period.

Follow-up of the grafted transduced cells will be performed on peripheral blood and bone marrow samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Fanconi Anemia complementation group A (FA-A)
* Minimum age 1 year
* Maximum age 21 years
* Lansky Index> 60%.
* Informed consent in accordance with current legal regulations.
* Number of cells to be transduced: At least 3x10^5 purified CD34+ / kg body weight.
* Negative result in the urine pregnancy test at the baseline visit for women of childbearing age, who should be committed to using an effective contraceptive method during the period of study participation.

Exclusion Criteria:

* Patients with an human leukocyte antigen (HLA) identical family donor.
* Evidence of myelodysplastic syndrome or leukemia, or cytogenetic abnormalities predicting the same in bone marrow aspirates. In this case, the studies carried out two months in advance of the patient's entry into the clinical trial will be considered valid.
* Evidence that the patient to be infused has signs of somatic mosaicism, with hematologic improvement.
* Any illness or concomitant process that in the opinion of the investigator incapacitates the subject for their participation in the study.
* Pre-existing sensory or motor impairment> = grade 2 according to the National Cancer Institute (NCl) criteria.
* Pregnant or lactating women.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to 3 years after infusion of transduced cells
  All adverse events will be registered for 3 years from infusion of transduced cells
Proportion of patients with at least 0.1 copy of the therapeutic vector per nucleated bone marrow or peripheral blood cells two years after infusion. | 2 years after infusion of transduced cells
  Detection of at least 0.1 copy of the therapeutic vector per nucleated bone marrow cell or peripheral blood cells two years after infusion.

SECONDARY OUTCOMES:
Proportion of patients with clinical hematological response after the infusion of autologous CD34 + cells transduced with the therapeutic lentiviral vector | 2 years after infusion of transduced cells
  Proportion of patients with clinical hematological response (improvement of cell blood counts at least in one hematological lineage).

CONTACTS AND LOCATIONS:
Overall Officials: Juan A Bueren, Study Director — CIEMAT/CIBERER/IIS.FJD
Locations (2):
- Spain (2):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Infantil del Niño Jesus, Madrid

REFERENCES:
- [Background] Adair JE, Sevilla J, Heredia CD, Becker PS, Kiem HP, Bueren J. Lessons Learned from Two Decades of Clinical Trial Experience in Gene Therapy for Fanconi Anemia. Curr Gene Ther. 2017;16(5):338-348. doi: 10.2174/1566523217666170119113029. PMID 28103787
- [Background] Molina-Estevez FJ, Nowrouzi A, Lozano ML, Galy A, Charrier S, von Kalle C, Guenechea G, Bueren JA, Schmidt M. Lentiviral-Mediated Gene Therapy in Fanconi Anemia-A Mice Reveals Long-Term Engraftment and Continuous Turnover of Corrected HSCs. Curr Gene Ther. 2015;15(6):550-62. doi: 10.2174/1566523215666150929110903. PMID 26415575
- [Background] Gonzalez-Murillo A, Lozano ML, Alvarez L, Jacome A, Almarza E, Navarro S, Segovia JC, Hanenberg H, Guenechea G, Bueren JA, Rio P. Development of lentiviral vectors with optimized transcriptional activity for the gene therapy of patients with Fanconi anemia. Hum Gene Ther. 2010 May;21(5):623-30. doi: 10.1089/hum.2009.141. PMID 20001454
- [Background] Jacome A, Navarro S, Rio P, Yanez RM, Gonzalez-Murillo A, Lozano ML, Lamana ML, Sevilla J, Olive T, Diaz-Heredia C, Badell I, Estella J, Madero L, Guenechea G, Casado J, Segovia JC, Bueren JA. Lentiviral-mediated genetic correction of hematopoietic and mesenchymal progenitor cells from Fanconi anemia patients. Mol Ther. 2009 Jun;17(6):1083-92. doi: 10.1038/mt.2009.26. Epub 2009 Mar 10. PMID 19277017
- [Background] Rio P, Navarro S, Guenechea G, Sanchez-Dominguez R, Lamana ML, Yanez R, Casado JA, Mehta PA, Pujol MR, Surralles J, Charrier S, Galy A, Segovia JC, Diaz de Heredia C, Sevilla J, Bueren JA. Engraftment and in vivo proliferation advantage of gene-corrected mobilized CD34+ cells from Fanconi anemia patients. Blood. 2017 Sep 28;130(13):1535-1542. doi: 10.1182/blood-2017-03-774174. Epub 2017 Aug 11. PMID 28801449
- [Result] Rio P, Navarro S, Wang W, Sanchez-Dominguez R, Pujol RM, Segovia JC, Bogliolo M, Merino E, Wu N, Salgado R, Lamana ML, Yanez RM, Casado JA, Gimenez Y, Roman-Rodriguez FJ, Alvarez L, Alberquilla O, Raimbault A, Guenechea G, Lozano ML, Cerrato L, Hernando M, Galvez E, Hladun R, Giralt I, Barquinero J, Galy A, Garcia de Andoin N, Lopez R, Catala A, Schwartz JD, Surralles J, Soulier J, Schmidt M, Diaz de Heredia C, Sevilla J, Bueren JA. Successful engraftment of gene-corrected hematopoietic stem cells in non-conditioned patients with Fanconi anemia. Nat Med. 2019 Sep;25(9):1396-1401. doi: 10.1038/s41591-019-0550-z. Epub 2019 Sep 9. PMID 31501599
- [Derived] Rio P, Zubicaray J, Navarro S, Galvez E, Sanchez-Dominguez R, Nicoletti E, Sebastian E, Rothe M, Pujol R, Bogliolo M, John-Neek P, Bastone AL, Schambach A, Wang W, Schmidt M, Larcher L, Segovia JC, Yanez RM, Alberquilla O, Diez B, Fernandez-Garcia M, Garcia-Garcia L, Ramirez M, Galy A, Lefrere F, Cavazzana M, Leblanc T, Garcia de Andoin N, Lopez-Almaraz R, Catala A, Barquinero J, Rodriguez-Perales S, Rao G, Surralles J, Soulier J, Diaz-de-Heredia C, Schwartz JD, Sevilla J, Bueren JA; FANCOLEN-1 gene therapy investigators. Haematopoietic gene therapy of non-conditioned patients with Fanconi anaemia-A: results from open-label phase 1/2 (FANCOLEN-1) and long-term clinical trials. Lancet. 2025 Dec 21;404(10471):2584-2592. doi: 10.1016/S0140-6736(24)01880-4. Epub 2024 Dec 3. PMID 39642902